CLINICAL TRIAL: NCT03897283
Title: Phase Ib Study of TQB2450 Combined With Anlotinib in Patients With Advanced Solid Tumors
Brief Title: Study of TQB2450 Combined With Anlotinib in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-Ib-04
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-03

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib + TQB2450 (Experimental): TQB2450 1200 milligrams (mg) administered intravenously (IV) on Day 1 of each 21-day cycle plus Anlotinib capsules given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Interventions: Drug: TQB2450; Drug: Anlotinib

INTERVENTIONS:
Drug: TQB2450 — TQB2450 1200 mg administered IV on Day 1 of each 21-day cycle
Drug: Anlotinib — Anlotinib capsules given orally in fasting conditions, dose ranging from 8 mg to 12 mg once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21). Initial dose is 10 mg. If there are no patients with DLT in first treatment cycle , begin to explore dose of 12 mg. If there are 2 or more patients in 3 patients with DLT, 8 mg dose is to explore.

SUMMARY:
TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1),which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors. As a novel multitarget tyrosine kinase inhibitor for tumor angiogenesis and proliferative signaling，anlotinib is approved for the treatment of patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) who have undergone progression or recurrence after ≥ 2 lines of systemic chemotherapy. The Phase III study showed that the Overall Survival (OS), Progression-Free Survival (PFS) and Overall Response Rate (ORR) were significantly better than placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced or metastatic solid tumor that is failure or absence of standard therapy with measurable lesion.
2. 18-70 years old；Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months.
3. The main organs function are normally, the following criteria are met:

   ① routine blood tests：hemoglobin (Hb) ≥ 90g/L (no blood transfusion and blood products within 14 days); absolute neutrophil count (ANC) ≥1.5×109/L; platelets (PLT) ≥ 100×109/L;

   ②Blood biochemical examination: alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN (when the liver is invaded，AST ≤ 5×ULN); total bilirubin (TBIL) ≤1.5×ULN (Gilbert syndrome patients，TBIL ≤ 3×ULN)；serum creatinine (Cr) ≤1.5×ULN，or calculated creatinine clearance (CrCl) ≥60 ml/min；

   ③Coagulation function: activated partial thromboplastin time (APTT) 、 international normalized ratio (INR) 、prothrombin time (PT) ≤1.5×ULN；

   ④ left ventricular ejection fraction (LVEF) measured by the Cardiac echocardiography ≥ 50%.
4. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization
5. Understood and signed an informed consent form.

Exclusion Criteria:

1. Prior therapy with anlotinib, anti-programmed cell death (PD)-1, anti-PD-L1 or other immunotherapy against PD-1/PD-L1.
2. Severe hypersensitivity occurs after administration of other monoclonal antibodies.
3. Has diagnosed and/or treated additional malignancy within 5 years prior to randomization. Exceptions include cured basal cell carcinoma of skin and carcinoma in situ of cervix.
4. Has any active autoimmune disease or history of autoimmune disease, such as autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis, asthma patients who need bronchiectasis for medical intervention; Subjects with the vitiligo without systemic treatment, psoriasis, alopecia, well-controlled type I diabetes mellitus, hypothyroidism stable on hormone replacement will not be excluded from this study.
5. Immunosuppressive therapy with immunosuppressive agents or systemic or absorbable local hormones (dosage > 10 mg/day prednisone or other therapeutic hormones) is required for the purpose of immunosuppression, and is still in use for 2 weeks after the first administration.
6. Has multiple factors affecting oral medication, such as inability to swallow, post-gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.
7. Has uncontrollable pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
8. Has spinal cord compression which was not cured or relieved through surgery and/or radiotherapy, or diagnosed spinal cord compression after treatment showed no clinical evidence of disease stabilization prior to randomization ≥1 week.
9. Has any bleeding or bleeding events ≥ grade 3 or with unhealed wounds, ulcerative , or fractures within 4 weeks prior to the first administration.
10. Has known central nervous system (CNS) metastases and/or carcinomatous meningitis. （subjects with treated brain metastases may participate provided the following criteria are met： Has no evidence of new or enlarging brain metastases at least two weeks after treatment of brain metastases ； Has stopped using corticosteroid before randomization, or used less than 10 mg prednisone or steady dose at least two weeks；If the patient is found to have active or new untreated or asymptomatic CNS metastases during the screening period, radiotherapy and/or operation for CNS metastatic lesion must be performed.
11. Has received chemotherapy, surgery, radiotherapy, the last treatment from the first dose less than 4 weeks, or oral targeted drugs for less than 5 half-lives, or oral fluorouracil pyridine drugs for less than 14 days, mitomycin C and nitrosourea for less than 6 weeks.
12. Has adverse events caused by previous therapy except alopecia that did not recover to ≤ grade 1.
13. Has major surgical procedure、biopsy or obvious traumatic injury within 28 days before randomization.
14. Has arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident including transient ischemic attack, deep vein thrombosis and pulmonary embolism.
15. Has drug abuse history that unable to abstain from or mental disorders.
16. Patients with any serious and/or uncontrollable disease, including :

    1. Has poor blood pressure control, systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 90 mmHg;
    2. Thrombotic events, ischemic attacks, myocardial infarction, grade 2 congestive heart failure or arrhythmias requiring treatment including QTc ≥ 480ms occurred within 6 months of first administration;
    3. Severe active or uncontrolled infections ≥ grade 2;
    4. Has known clinical history of liver diseases, including viral hepatitis, known carriers of hepatitis B virus (HBV) must exclude active HBV infection, that is, HBV DNA positive > 1 *104 copies/mL or > 2000 IU/mL, known hepatitis C virus infection (HCV) and HCV RNA positive > 1 *103 copies/mL, or other decompensated hepatitis and chronic hepatitis, which require antiviral treatment;
    5. HIV positive;
    6. Poor control of diabetes mellitus, fasting blood-glucose ≥ grade 2;
    7. Urinary routine indicated that urinary protein ≥ ++ and confirmed 24-hour urinary protein quantification > 1.0 g.
17. Has vaccinated with vaccines or attenuated vaccines within 4 weeks prior to first administration.
18. Has participated in other anticancer drug clinical trials within 4 weeks.
19. According to the judgement of the researchers, there are other factors that may lead to the termination of the study. For example, other serious diseases including mental disorders need to be treated together, serious laboratory abnormalities, accompanied by family or social factors, which will affect the safety of the subjects, or the collection of data and samples.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 21 days
  DLT defined as any of the following events occurring during the study related to drugs : （1） ≥grade 3 non-hematologic toxicity, except for the following conditions: Nausea, vomiting, diarrhea, constipation, electrolyte imbalance that downgrade within 1 week after supportive treatment； Grade 3 fatigue ≤ 7 days duration； Grade 3 hypertension that can be controlled within 1 week by medication； Alopecia, fever caused by tumor or infection, and elevated alkaline phosphatase; （2）Grade 4 neutropenia, thrombocytopenia, and hemoglobin reduction confirmed by at least 2 tests within 2 days; Grade 3 thrombocytopenia with bleeding tendency confirmed by at least 2 tests within 2 days; （3）Grade 3 neutropenia with fever confirmed at least 2 times within 2 days (neutrophil count <1.0×109 / L; fever ≥38.5℃) （4）Immune-related interstitial pneumonia ≥ grade 2 ； （5）Decreased ventricular ejection fraction ≥ grade 2 ； （6）Retinal vein occlusion (RVO), uveitis ≥ grade 2 , and other more serious ocular
Maximum tolerated dose (MTD) | Baseline up to 21 days
  MTD defined as the highest dose level at which less than or equal to 2 of 6 subjects experience dose limiting toxicity (DLT)
Determine the Recommended Phase II Dose (RP2D) | Up to approximately 18 months
  The RP2D defined as the lower dose level to MTD based on the safety profile

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 18 months
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR)
Disease control rate (DCR) | Up to approximately 18 months
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD)
Progression-free survival (PFS) | Up to approximately 18 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause
Overall survival (OS) | Up to approximately 24 months
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive
Adverse Event: Drug dose adjustment | up to approximately 18 months
  Security Index

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin Cancer Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No